CLINICAL TRIAL: NCT01454193
Title: Are we Loading Our Patients With Sodium During Hemodialysis Treatments?
Status: Completed | Type: Observational
Sponsor: Renal Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 078-08
Record Dates: First submitted 2011-10-13; First posted 2011-10-18 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objectives of the data search is to find out if there is correlation between pre, post serum sodium concentration, dialysate sodium concentration, interdialytic weight gain and associated changes in pre and post systolic and diastolic blood pressure, mean arterial pressure, number of blood pressure medications and adherence to 3 times per week dialysis, mortality.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patient

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients at Renal Research Institute and Fresenius clinics
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2001-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kotanko, MD, Principal Investigator — Renal Research Institute
Locations (1):
- Renal Research Institute, New York, New York, United States